CLINICAL TRIAL: NCT05391191
Title: Prospective Clinical Study on the Safety and Clinical Feasibility of Exploring TRISKELE® Transcatheter Aortic Valve System in the Treatment of Severe Aortic Stenosis
Brief Title: Safety and Feasibility of TRISKELE in Severe AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRISKELE
Record Dates: First submitted 2022-05-22; First posted 2022-05-25 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MitrAssist TRISKELE® transcatheter aortic valve system (Experimental): Device: MitrAssist TRISKELE® transcatheter aortic valve system
  Interventions: Device: MitrAssist TRISKELE® transcatheter aortic valve system

INTERVENTIONS:
Device: MitrAssist TRISKELE® transcatheter aortic valve system — Patients were treated with MitrAssist TRISKELE® transcatheter aortic valve system

SUMMARY:
This clinical study is a prospective、single arm and exploratory study, to explore the feasibility and safety of MitrAssist TRISKELE® transcatheter aortic valve system in the treatment of patients with severe aortic stenosis.

DETAILED DESCRIPTION:
This study was a prospective、single arm clinical trial design. For patients with surgical contraindications or high-risk symptomatic severe aortic stenosis, MitrAssist TRISKELE® transcatheter aortic valve system was performed by aortic valve replacement. Patients were followed up 30 days (± 7 days) after operation for the feasibility and safety analysis to explore the test device in patients with surgical contraindications or high-risk symptomatic severe aortic stenosis.In this study, a clinical trial institution meeting the national qualification is planned to be selected as the clinical research center, and 7 patients are planned to be selected.

The success rate of operation 30 days after operation was taken as the main evaluation index and the success of device implantation, the result of echocardiography evaluation of valve function, the improvement rate of NYHA cardiac function classification, six minute walking distance and the score of Kansas City Cardiomyopathy Questionnaire were taken as the secondary evaluation indexes, to evaluate clinical effectiveness of TRISKELE® transcatheter aortic valve system; Adverse events, serious adverse events, major cardiovascular and cerebrovascular adverse events, device defects, vital signs and laboratory examination results were used as safety indicators to evaluate the safety of the test device .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years old;
2. Patients with symptomatic severe aortic stenosis (echocardiographic mean pressure gradient across aortic valve ≥ 40mmhg, or blood flow velocity across aortic valve ≥ 4.0m/s, or aortic valve area < 0.8cm2, or effective aortic valve area index < 0.5cm2/m2);
3. Patients with biological valve decay meeting the criteria in (2) above;
4. NYHA grade ≥ grade II;
5. The life expectancy after artificial valve implantation is more than 1 year;
6. Patients who are anatomically suitable for transcatheter aortic valve implantation;
7. Two or more cardiothoracic surgeons evaluate and record it as surgical contraindication or as high-risk surgery and unsuitable for routine surgery;
8. Patients who can understand the purpose of the trial, voluntarily participate in and sign informed consent, and are willing to accept relevant examination and clinical follow-up.

Exclusion Criteria:

1. Acute myocardial infarction occurred within 30 days before this treatment (WHO definition: Q-wave MI, or non-Q-wave MI with elevated creatine kinase isoenzyme and troponin T);
2. Patients whose aortic root anatomy and lesions are not suitable for artificial valve implantation;
3. Compound aortic valve disease (aortic stenosis with severe regurgitation); Severe mitral regurgitation;
4. Hematological malignancies, hemophilia and other coagulation disorders;
5. Hemodynamic instability, requiring mechanical cardiac assistance;
6. Emergency operation for any reason;
7. Obstructive hypertrophic cardiomyopathy;
8. Severe left ventricular dysfunction, left ventricular ejection fraction (LVEF) < 30%;
9. Severe right ventricular dysfunction;
10. Echocardiography showed the presence of intracardiac mass, thrombus or vegetations;
11. Active peptic ulcer or upper gastrointestinal hemorrhage within 3 months;
12. Allergic to nickel titanium alloy, stainless steel alloy, PU (polyurethane), or contrast agent; Unable to tolerate anticoagulant and antiplatelet therapy;
13. Cerebrovascular events (CVA) occurred within 3 months, including ischemic stroke and hemorrhagic stroke, excluding transient ischemic attack (TIA);
14. Vascular diseases affecting the instrument approach;
15. Infective endocarditis in active phase or other active infections;
16. Those who have participated in clinical trials of other drugs or medical devices before enrollment and have not reached the time limit of the main research endpoint.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Technical success | at exit from procedure room
  Freedom from mortality; Successful access, delivery of the device, and retrieval of the delivery System; Correct positioning of a single prosthetic heart valve into the proper anatomical location; Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Device success | within 30 days after operation
  Technical success; Freedom from mortality; Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication; Intended performance of the valve (mean gradient <20 mmHg, peak velocity<3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation)

SECONDARY OUTCOMES:
Early safety endpoint | within 30 days after operation
  Freedom from all-cause mortality; Freedom from all stroke; Freedom from VARC type 2-4 bleeding (in trials where control group is surgery, it is appropriate to include only Type 3 and 4 bleeding); Freedom from major vascular, access-related, or cardiac structural complication; Freedom from acute kidney injury stage 3 or 4; Freedom from moderate or severe aortic regurgitation; Freedom from new permanent pacemaker due to procedure-related conduction abnormalities; Freedom from surgery or intervention related to the device
six minute walk distance (6MWD) test | within 30 days after operation
  The six minute walk distance (6MWD) test (see Appendix II) was used to record the patients' six minute walk distance before operation and 30 days after operation. The six minute walk test is mainly used to evaluate the efficacy of treatment intervention in patients with moderate and severe cardiovascular diseases, and can objectively reflect the actual daily activity ability
The quality of life improved 30 days after operation | within 30 days after operation
  SF-12 quality of life table was used to score the cardiac function improvement before discharge and 30 days after operation. NYHA classification scheme was adopted for the classification of cardiac function.

CONTACTS AND LOCATIONS:
Overall Officials: JUNBO GE, PHD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hopital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No